CLINICAL TRIAL: NCT03228498
Title: Pilot Study on the Association Choline Alphoscerate-Nimodipine in Patients With Subcortical Vascular Cognitive Impairment
Brief Title: Choline Alphoscerate-Nimodipine in Vascular Cognitive Impairment
Acronym: CONIVAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Collaborators: MDM S.p.A. (Other)
Responsible Party: Principal Investigator, Leonardo Pantoni, Professor, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-003188-13
Record Dates: First submitted 2017-07-19; First posted 2017-07-25 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Vascular Cognitive Impairment
MeSH Terms: interventions — Glycerylphosphorylcholine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind (Participant, Investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Choline alphoscerate (Experimental): Drug: Choline alphoscerate 1200 mg per day and Nimodipine 90 mg per day
  concomitant administration
  Interventions: Drug: Choline alphoscerate
- Placebo (Placebo Comparator): Placebo and Drug: Nimodipine 90 mg per day only
  concomitant administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Choline alphoscerate — Choline alphoscerate 600 mg b.i.d plus Nimodipine 30 mg t.i.d
  Other Names: Delecit
  Arms: Choline alphoscerate
Drug: Placebo — Placebo b.i.d plus Nimodipine 30 mg t.i.d
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether the combination of choline alphoscerate 1200mg per day and nimodipine 90mg per day given orally is more effective than the combination nimodipine placebo in reducing cognitive decline in patients with subcortical vascular cognitive impairment

DETAILED DESCRIPTION:
Cerebrovascular diseases represent the second most common cause of dementia after Alzheimer's disease. Since cerebrovascular diseases are age-related, an increase in the incidence of this pathology, due to the aging of the population, is expected.

Vascular cognitive impairment (VCI) embraces a broad-spectrum of cognitive disorders related to cerebrovascular diseases, from mild cognitive impairment to severe dementia. VCI is an extremely disabling condition with severe consequences in terms of direct (e.g., clinic visits, prescriptions, hospital accesses, etc..) and indirect costs (e.g., loss of patient's and caregiver's productivity, consequent increase in psychological burdens, etc.).

The two main categories of VCI include post-stroke dementia and vascular cognitive impairment caused by cerebral small vessel disease. Given its great weight in the dementia field, the interest of the international scientific community is currently focused on small vessel disease, its neuroradiological definition and its clinical consequences.

Despite these relevant facts, there are no approved therapies for VCI due to small disease.

In the past, several drugs have been tested in patients affected by VCI with variable results. A large amount of data come from studies performed with drugs approved for the treatment of Alzheimer's disease (such as acetylcholinesterase inhibitors, N-methyl-D-aspartate glutamate receptor antagonists, cholinergic precursors, calcium-channel blockers).

Choline alphoscerate and nimodipine have demonstrated some positive effects in VCI patients, and a confirmation of this effect in quantitative terms could permit to obtain the prescribing license for VCI.

It may be possible that a combined treatment with two drugs that act on different targets could achieve better results in patients affected by subcortical VCI, also in consideration of the fact that small vessel disease is characterized by a damage of microvessels and produces a cortical disconnection.

The main objective of this study is to assess whether the combination of choline alphoscerate 1200mg per day and nimodipine 90mg per day given orally is more effective than the combination of nimodipine and placebo in reducing cognitive decline in patients with subcortical VCI.

Project design:

The present study is a 2-year prospective, double-blinded, randomized trial. The enrolment will be carried out at Vascular Cognitive (VASCOG) clinic of the Careggi University Hospital in Florence, Italy. Sixty-eight patients will be enrolled according to the following inclusion criteria: 1) Cognitive impairment of mild to moderate degree defined by a Clinical Deterioration Rating (CDR) score range between 0.5 and 2.0; 2) Evidence on brain MRI of white matter hyperintensities (leukoaraiosis of moderate or severe degree according to the modified Fazekas visual scale and/or presence of lacunar infarcts); 3) Consent to participation in the study.

All enrolled patients will be evaluated at baseline according to the study protocol that includes: 1) Clinical assessment; 2) Functional, quality of life and mood assessments; 3) Extensive neuropsychological evaluation.

After baseline assessment, participants will be randomly assigned to one of two arms of treatment: 1) nimodipine 90 mg/die t.i.d plus placebo b.i.d; 2) nimodipine 90 mg t.i.d plus choline alphoscerate 1200 mg/die b.i.d. Treatment will be given for a total of 12 months.

Each patient will be followed-up at 6 and 12 months after baseline. During the first follow-up visit, clinical assessment and evaluation of side effects and compliance to treatment will be carried out; during the second follow up visit, clinical assessment, an extensive neuropsychological evaluation, and mood, functional, and quality of life assessments will be performed according to the baseline protocol.

The primary end point of this study is to assess the cognitive decline, expressed as the loss of at least 2 points on the Montreal Cognitive Assessment (MoCA) test 12 months after baseline. A comparative analysis of MoCA test values between two groups will be assessed by covariate analysis (ANCOVA) introducing in the statistical model these two covariates: arm of treatment and MoCA test score at the baseline (based on the exploratory nature of this study the significance level on the covariate arm of treatment is 20%).

ELIGIBILITY:
Inclusion Criteria:

1. Cognitive impairment from mild to moderate degree defined by a Clinical Deterioration Rating (CDR) score range between 0.5 and 2.0.
2. Evidence on brain MRI of white matter hyperintensities (leukoaraiosis of moderate or severe degree according to the modified Fazekas visual scale and/or presence of lacunar infarcts).
3. Consent to participation in the study.

Exclusion Criteria:

1. Absence of objectionable cognitive impairment or presence of dementia of severe degree defined by CDR score > 2.0.
2. Unavailability of brain MRI (in case of absolute contraindications, the use of cranial CT is allowed).
3. Expected poor compliance with the study protocol.
4. Past diagnosis of major depression, schizophrenia, major anxiety syndrome, or manic- depressive illness.
5. Diagnosis of degenerative cognitive impairment based on clinical and/or neuroradiological findings (i.e., patients with prevailing memory impairment, or with medial temporal atrophy on brain MRI in absence of evident vascular abnormalities; i.e., Alzheimer disease as defined using the National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association criteria, Parkinson disease, Huntington disease, frontotemporal dementia).
6. Diagnosis of cognitive impairment from other causes (i.e., vitamine B12 and folic acid deficiency, thyroid disorders, metabolic diseases, head trauma, tumor or infections of the central nervous system, normal pressure hydrocephalus).
7. Medical conditions expected to progress, recur, or change to such a degree to interfere with the assessment of the clinical and mental status.
8. Clinically relevant cardiac or pulmonary insufficiency.
9. Relevant electrocardiograph abnormalities; bradycardia (50 bpm) or tachycardia (120 bpm) under resting conditions.
10. Myocardial infarction within the past 6 months.
11. Stroke still requiring neurological rehabilitation.
12. Severe/untreated blood pressure (systolic 180 mm Hg, diastolic 95 mm Hg).
13. Clinically relevant liver function impairment.
14. Insulin-dependent diabetes mellitus.
15. Idiopathic epilepsy and anti-epileptic treatment.
16. Severe anemia (Hb <10 mg/dL).
17. Severe gastrointestinal disease.
18. Cancer.
19. Known intolerance to study drugs.
20. Coexistent serious illnesses that would imply a drop-out before the end of the trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Cognitive decline evaluated by the change of MoCA test score compared with Baseline | 12 months
  Cognitive decline: expressed as the loss of at least 2 points on Montreal Cognitive Assessment (MoCA) test

SECONDARY OUTCOMES:
Evaluation of selective attention | 12 months
  Selective attention assessed by means of Color Word Stroop Test (CWST)
Evaluation of divided attention | 12 months
  Divided attention assessed by means of Trail Making Test (TMT)
Evaluation of maintained attention | 12 months
  Maintained attention assessed by means of Symbol Digit Modalities Test (SDMT)
Evaluation of memory | 12 months
  Memory assessed by means of Rey Auditory-Verbal Learning Test (RAVLT)
Assessment of functional status | 12 months
  Functional status measured by Disability Assessment for Dementia scale (DAD)
Evaluation of depressive symptoms | 12 months
  Depressive symptoms assessed by means of Center for Epidemiological Studies Depression scale (CES-D)
Assessment of quality of life | 12 months
  Quality of life assessed by means of Stroke-Adapted Sickness Impact Profile (SA-SIP30)
Assessment of drugs' safety and tolerability. | 12 months
  Evaluation of drugs' side effects incidence between two groups of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Stroke Unit, VAS-COG clinic, Azienda Ospedaliero Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Brien JT, Erkinjuntti T, Reisberg B, Roman G, Sawada T, Pantoni L, Bowler JV, Ballard C, DeCarli C, Gorelick PB, Rockwood K, Burns A, Gauthier S, DeKosky ST. Vascular cognitive impairment. Lancet Neurol. 2003 Feb;2(2):89-98. doi: 10.1016/s1474-4422(03)00305-3. PMID 12849265
- [Background] Pantoni L. Cerebral small vessel disease: from pathogenesis and clinical characteristics to therapeutic challenges. Lancet Neurol. 2010 Jul;9(7):689-701. doi: 10.1016/S1474-4422(10)70104-6. PMID 20610345
- [Background] Wardlaw JM, Smith C, Dichgans M. Mechanisms of sporadic cerebral small vessel disease: insights from neuroimaging. Lancet Neurol. 2013 May;12(5):483-97. doi: 10.1016/S1474-4422(13)70060-7. PMID 23602162
- [Background] Wardlaw JM, Smith EE, Biessels GJ, Cordonnier C, Fazekas F, Frayne R, Lindley RI, O'Brien JT, Barkhof F, Benavente OR, Black SE, Brayne C, Breteler M, Chabriat H, Decarli C, de Leeuw FE, Doubal F, Duering M, Fox NC, Greenberg S, Hachinski V, Kilimann I, Mok V, Oostenbrugge Rv, Pantoni L, Speck O, Stephan BC, Teipel S, Viswanathan A, Werring D, Chen C, Smith C, van Buchem M, Norrving B, Gorelick PB, Dichgans M; STandards for ReportIng Vascular changes on nEuroimaging (STRIVE v1). Neuroimaging standards for research into small vessel disease and its contribution to ageing and neurodegeneration. Lancet Neurol. 2013 Aug;12(8):822-38. doi: 10.1016/S1474-4422(13)70124-8. PMID 23867200
- [Background] Pantoni L. Treatment of vascular dementia: evidence from trials with non-cholinergic drugs. J Neurol Sci. 2004 Nov 15;226(1-2):67-70. doi: 10.1016/j.jns.2004.09.014. PMID 15537523
- [Background] Smith EE, Cieslak A, Barber P, Chen J, Chen YW, Donnini I, Edwards JD, Frayne R, Field TS, Hegedus J, Hanganu V, Ismail Z, Kanji J, Nakajima M, Noor R, Peca S, Sahlas D, Sharma M, Sposato LA, Swartz RH, Zerna C, Black SE, Hachinski V. Therapeutic Strategies and Drug Development for Vascular Cognitive Impairment. J Am Heart Assoc. 2017 May 5;6(5):e005568. doi: 10.1161/JAHA.117.005568. No abstract available. PMID 28476873
- [Background] Di Perri R, Coppola G, Ambrosio LA, Grasso A, Puca FM, Rizzo M. A multicentre trial to evaluate the efficacy and tolerability of alpha-glycerylphosphorylcholine versus cytosine diphosphocholine in patients with vascular dementia. J Int Med Res. 1991 Jul-Aug;19(4):330-41. doi: 10.1177/030006059101900406. PMID 1916007
- [Background] Pantoni L, Carosi M, Amigoni S, Mascalchi M, Inzitari D. A preliminary open trial with nimodipine in patients with cognitive impairment and leukoaraiosis. Clin Neuropharmacol. 1996 Dec;19(6):497-506. doi: 10.1097/00002826-199619060-00003. PMID 8937788
- [Background] Pantoni L, del Ser T, Soglian AG, Amigoni S, Spadari G, Binelli D, Inzitari D. Efficacy and safety of nimodipine in subcortical vascular dementia: a randomized placebo-controlled trial. Stroke. 2005 Mar;36(3):619-24. doi: 10.1161/01.STR.0000155686.73908.3e. Epub 2005 Feb 3. PMID 15692125
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Poggesi A, Salvadori E, Pantoni L, Pracucci G, Cesari F, Chiti A, Ciolli L, Cosottini M, Del Bene A, De Stefano N, Diciotti S, Dotti MT, Ginestroni A, Giusti B, Gori AM, Nannucci S, Orlandi G, Pescini F, Valenti R, Abbate R, Federico A, Mascalchi M, Murri L, Inzitari D. Risk and Determinants of Dementia in Patients with Mild Cognitive Impairment and Brain Subcortical Vascular Changes: A Study of Clinical, Neuroimaging, and Biological Markers-The VMCI-Tuscany Study: Rationale, Design, and Methodology. Int J Alzheimers Dis. 2012;2012:608013. doi: 10.1155/2012/608013. Epub 2012 Apr 8. PMID 22550606
- [Derived] Salvadori E, Poggesi A, Donnini I, Rinnoci V, Chiti G, Squitieri M, Tudisco L, Fierini F, Melone A, Pescini F, Pantoni L. Efficacy and Safety of the Association of Nimodipine and Choline Alphoscerate in the Treatment of Cognitive Impairment in Patients with Cerebral Small Vessel Disease. The CONIVaD Trial. Drugs Aging. 2021 Jun;38(6):481-491. doi: 10.1007/s40266-021-00852-8. Epub 2021 Apr 15. PMID 33855653
- [Derived] Salvadori E, Poggesi A, Donnini I, Rinnoci V, Chiti G, Squitieri M, Tudisco L, Fierini F, Melone A, Pescini F, Pantoni L. Association of nimodipine and choline alphoscerate in the treatment of cognitive impairment in patients with cerebral small vessel disease: study protocol for a randomized placebo-controlled trial-the CONIVaD trial. Aging Clin Exp Res. 2020 Mar;32(3):449-457. doi: 10.1007/s40520-019-01229-z. Epub 2019 May 30. PMID 31148099